CLINICAL TRIAL: NCT00808587
Title: Scripps Genomics Health Initiative
Status: Active, not recruiting | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: Navigenics, Inc. (Industry); Affymetrix, Inc. (Industry)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Scripps Translational Science Institute
Other Study IDs: HSC# 08-5069
Record Dates: First submitted 2008-12-09; First posted 2008-12-16 (Estimated); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Genes
Keywords: Genomic Scan; Personalized Medicine; Gene testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No Treatment

SUMMARY:
The specific aims for this project are to enroll up to 10,000 subjects who will have their genomes surveyed using the Navigenics™ Health Compass technology. The Navigenics Health Compass helps you understand what your genetic variants have to say about the future of your health, and gives you action steps to take control of your health today. In addition, the investigators will assess how the Navigenics Health Compass, results affect lifestyle decisions. The phenotyping information that can be analyzed with the resulting Navigenics genotype information will assist in identifying genetic variations associated with other traits and diseases.

The uses of molecular markers such as cholesterol and glucose levels to assess disease risk are well established in clinical medicine today. Although these tools are useful in screening for subclinical disease, their predictive value is limited. Until recently, these molecular markers were the best risk assessment and screening tools in existence. Since the completion of the Human Genome Project, the era of personalized medicine, which exploits knowledge of the genes an individual carries that may predispose him/her to disease, has come to the forefront of research.

The Navigenics Health Compass technology assesses risk for about over 20 common diseases and provides subjects with more accurate assessments of their individual predictive risk for developing these conditions than traditional biomarkers such as cholesterol and glucose levels. This may positively influence changes in lifestyle, as well as decisions to seek further medical evaluation associated with preventive strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Able to read, write, and fluently understand English.
* Be reliable, cooperative, and willing to comply with all protocol specified procedures.
* Be able to understand and grant informed consent.
* Be able to provide payment for services rendered.
* Have an email address.

Exclusion Criteria:

* Intake of anything orally, i.e., food, beverage, cigarettes, brushing of teeth, 30 minutes prior to providing saliva sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Scripps Health employees, friends, family, and the general population
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be lifestyle changes based on the subject's genetic risk(s). | Three and 12 months

SECONDARY OUTCOMES:
The secondary endpoint will be to evaluate the frequency of subjects changing their lifestyle based on factors such as education, gender, disease history, and related items. | Three and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric J. Topol, MD, Principal Investigator — Scripps Translational Science Institute
Locations (1):
- Scripps Health, San Diego, California, United States

REFERENCES:
- See also: Scripps Genomic Health Initiative — http://www.stsiweb.org/index.php/support/scripps_genomic_health_initiative/